CLINICAL TRIAL: NCT05374798
Title: Using Wearable Technology to Develop Biomarker-Driven Intervention for Alcohol-Facilitated Intimate Partner Violence
Brief Title: Wearable Technology and Alcohol-Facilitated Intimate Partner Violence
Acronym: START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Julianne Flanagan, Associate Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00116875; R21AA029235 (NIH)
Record Dates: First submitted 2022-04-14; First posted 2022-05-16 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Abuse; IPV; Couples
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Participants will wear activity trackers (Garmin smartwatch) equipped with continuous ambulatory physiological monitoring and geolocation. Ecological momentary assessment (EMA; 4 times daily plus optional event-triggered reports) of alcohol use, couple conflict including IPV, and affect will be completed via smartphone application for 28 days. During days 21-28, participants will also be prompted to complete a 10 minute self-administered HRV-B session at least once daily. Subjective usability, feasibility, and acceptability of HRV-B will be assessed The investigative team is not testing the Garmin smartwatch, but the use of EMA and HRV biofeedback as a mechanism to modulate alcohol use and IPV among couples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart Rate Variability-Biofeedback via Smartwatch Device Intervention (Experimental): Participants will wear activity trackers equipped with continuous ambulatory physiological monitoring and geolocation. Ecological momentary assessment (EMA; 4 times daily plus optional event-triggered reports) of alcohol use, couple conflict including IPV, and affect will be completed via smartphone application for 28 days. During days 21-28, participants will also be prompted to complete a 10 minute self-administered HRV-B session at least once daily. Subjective usability, feasibility, and acceptability of HRV-B will be assessed.
  Interventions: Device: Heart Rate Variability-Biofeedback (HRV-B) via Smartwatch Device Intervention

INTERVENTIONS:
Device: Heart Rate Variability-Biofeedback (HRV-B) via Smartwatch Device Intervention — Participants will wear activity trackers equipped with continuous ambulatory physiological monitoring and geolocation. Ecological momentary assessment (EMA; 4 times daily plus optional event-triggered reports) of alcohol use, couple conflict including IPV, and affect will be completed via smartphone application for 28 days. During days 21-28, participants will also be prompted to complete a 10 minute self-administered HRV-B session at least once daily. Subjective usability, feasibility, and acceptability of HRV-B will be assessed. HRV-B will guide participants in an evidence-based paced breathing technique (about 6 breaths per minutes) using visualization on thier mobile device of thier real-time respiratory and cardiac parameters.
  During days 21-28, participants will also be prompted to complete a 10 minute self-administered HRV-B session at least once daily. Subjective usability, feasibility, and acceptability of HRV-B will be assessed.

SUMMARY:
This project seeks to develop interactive treatment options to successfully reduce AUD and IPV concurrently. The purpose of the study is to examine the usability, feasibility, and acceptability of wearable activity trackers (like a smart watch) and use of a cell phone application (app) among couples. The investigators are also testing the use of this device and app will affect alcohol use and couple conflict.

This study involves a screening phase and a 28 observation period where participants are asked to wear a smart watch, complete assessments and provide feedback.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) and acute alcohol intoxication are well-established precipitants of intimate partner violence (IPV). Approximately one third of U.S. adults experience IPV during their lifetimes. Recent data indicate that IPV negatively impacts AUD treatment and increases risk of relapse. Although behavioral treatments targeting AUD and IPV are effective for some women and men, efficacy is commonly limited by high dropout rates, poor working alliance, and low readiness to change. As a result, there is a critical and persistent need to develop dynamic treatment options to successfully reduce AUD and IPV concurrently.

Mitigating maladaptive physiological reactivity in the form of respiratory sinus arrhythmia measure of heart rate variability (HRV) is one promising pathway to achieve this goal. HRV is an autonomic biomarker of arousal relevant to AUD pathophysiology, alcohol consumption, and treatment outcomes. HRV is also an emerging mechanism underlying alcohol-facilitated IPV. Growing evidence suggests that biofeedback interventions to modulate physiological, emotional, and behavioral stress responses are feasible, acceptable, and may reduce AUD symptoms such as craving to improve long-term AUD recovery. This data suggests that remote, self-administered biofeedback interventions hold promise as a discreet, accessible and low cost standalone or adjunct treatment option for AUD patients with high risk behaviors such as IPV. Thus, the primary objective of the proposed project is to use wearable technology to develop proof-of-concept of HRV as a biomarker of alcohol-facilitated IPV in naturalistic settings. The secondary objective is to examine the preliminary usability, feasibility, and acceptability of a remote, self-administered HRV-B intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Any gender identity; any race or ethnicity; any sexual orientation; aged 21-70 years.
2. Married, cohabiting, or in a committed relationship for ≥ 6 months.
3. English fluency and cognitive functioning sufficient to provide informed consent and participate accurately (score ≥ 26 on the Mini-Mental Status Exam [MMSE]).
4. At least one partner within each dyad must meet DSM-V diagnostic criteria for current AUD (assessed by the QuickSCID) and consume ≥ 2 hazardous drinking episodes (i.e., 4 or more drinks for women, 5 or more for men in ≤ 2 hours) per month in the past three months.
5. At least one partner within each dyad must endorse ≥1 instance of IPV with their current partner in the past 6 months (assessed by the Revised Conflict Tactics Scale [CTS-2]).
6. Maintenance of psychotropic medications on a stable dose for at least 4 weeks before study initiation.

Exclusion Criteria:

1. Meeting DSM-5 criteria for a history of or current psychotic or bipolar disorders.
2. Meeting DSM-5 diagnostic criteria for moderate or severe drug use disorder (e.g., cannabis). Concurrent mild drug use disorders are acceptable due to the marked co-occurrence in AUD populations.
3. Alcohol withdrawal as indicated by CIWA-Ar scores >8.
4. Current suicidal or homicidal ideation and intent.
5. Serious cardiovascular health conditions (e.g., pacemaker, cardiac arrhythmia, hypertension) because the safety of HRV-B has not yet been established in these populations.
6. Treatment on medications such as lithium, methadone, alpha or beta blockers or cholinergic/ anticholinergic medications likely to confound normative cardiovascular responding.
7. Current neurologic conditions or history of traumatic brain injury.
8. Severe and unilateral IPV in the past 6 months.
9. Current pregnancy.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Addiction Sciences Division-Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through internet advertisements, clinician referrals and community providers, flyers, and from prior research studies. Following preliminary eligibility screening, couples completed private written informed consent and a baseline assessment separately for privacy. The baseline assessment included a alcohol and drug screen, battery of standardized self-report and interview measures. Recruitment and enrollment occurred from November 2022 through April 2024.
Pre-assignment Details: Participants were N=46 couples (N=92 individuals) where at least one partner within each dyad must have 1) met Diagnostic and Statistical Manual of Mental Disorders (DSM-V) diagnostic criteria for current alcohol use disorder and current alcohol use, and 2) have reported at least one instance of physical intimate partner violence in the past two years.
Groups:
- Full Sample: Participants were N=46 couples (N=92 individuals) with current alcohol use disorder and recent physical intimate partner violence (IPV). All participants completed 28 days of ecological momentary assessment (EMA) (4 times daily plus optional event-driven reports) of alcohol use, couple conflict including IPV, and affect via smartphone.
Period: Overall Study
Arm/Group | Full Sample
Started (N=92 participants (N=46 couples)) | 92 (N=92 individual participants)
Completed (N=86 participants (N=43 couples).N is represented as individuals in order to accurately account for those who did not complete the study. N=2 individuals were lost to follow up. N=2 individuals withdrew from the study and N=2 were withdrawn by the principal investigator (partners remained enrolled).) | 86 (N=86 individual participants)
Not Completed | 6
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2
Not completed — Withdrawn by Principal Investigator. | 2

BASELINE CHARACTERISTICS:
Population: The full sample consists of N=92 participants. Outcome measures were collected and reported on N=86 participants (2 participants dropped out, 2 participants were lost to follow up and 2 participants were withdrawn by Principal Investigator).
Groups:
- Full Sample: Participants were N=46 couples with current alcohol use disorder (AUD) and recent physical intimate partner violence (IPV). All participants completed 28 days of ecological momentary assessment (EMA); 4 times daily plus optional event-driven reports) of alcohol use, couple conflict including IPV, and affect via smartphone.
Arm/Group | Full Sample
Number analyzed (Participants) | 92
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Identified Patient and Partner listed in individual rows.
  years
    Total Sample | 36.8 (9.7)
    Identified Patient: number analyzed (Participants) | 46
    Identified Patient | 37.0 (10.1)
    Partner: number analyzed (Participants) | 46
    Partner | 36.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Identified Patient and Partner listed in individual rows.
  Participants
    Total Sample: Female | 52
    Total Sample: Male | 40
    Identified Patient: number analyzed (Participants) | 46
    Identified Patient: Female | 22
    Identified Patient: Male | 24
    Partner: number analyzed (Participants) | 46
    Partner: Female | 30
    Partner: Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Identified Patient and Partner listed in individual rows.
  Participants
    Total Sample: Hispanic or Latino | 11
    Total Sample: Not Hispanic or Latino | 81
    Total Sample: Unknown or Not Reported | 0
    Identified Patient: number analyzed (Participants) | 46
    Identified Patient: Hispanic or Latino | 6
    Identified Patient: Not Hispanic or Latino | 40
    Identified Patient: Unknown or Not Reported | 0
    Partner: number analyzed (Participants) | 46
    Partner: Hispanic or Latino | 5
    Partner: Not Hispanic or Latino | 41
    Partner: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Identified Patient and Partner listed in individual rows.
  Participants
    Total Sample: American Indian or Alaska Native | 1
    Total Sample: Asian | 4
    Total Sample: Native Hawaiian or Other Pacific Islander | 1
    Total Sample: Black or African American | 31
    Total Sample: White | 48
    Total Sample: More than one race | 7
    Total Sample: Unknown or Not Reported | 0
    Identified Patient: number analyzed (Participants) | 46
    Identified Patient: American Indian or Alaska Native | 1
    Identified Patient: Asian | 2
    Identified Patient: Native Hawaiian or Other Pacific Islander | 1
    Identified Patient: Black or African American | 15
    Identified Patient: White | 23
    Identified Patient: More than one race | 4
    Identified Patient: Unknown or Not Reported | 0
    Partner: number analyzed (Participants) | 46
    Partner: American Indian or Alaska Native | 0
    Partner: Asian | 2
    Partner: Native Hawaiian or Other Pacific Islander | 0
    Partner: Black or African American | 16
    Partner: White | 25
    Partner: More than one race | 3
    Partner: Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 92

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate Variability During Alcohol-Facilitated Intimate Partner Violence (IPV)
Description: Heart Rate Variability (HRV) was measured by Respiratory Sinus Arrhythmia (RSA) data derived from Garmin smart watch. RSA is a type/contributor of HRV that occurs when the heart rate changes with normal breathing (measure of changes in time in between heartbeats). RSA is an autonomic biomarker of arousal relevant to AUD pathophysiology. Alcohol-facilitated intimate partner violence (IPV) was measured by the self-reported presence of alcohol use, IPV or conflict on ecological momentary assessments (EMA; 4 times daily plus optional event-daily or event-driven) via a smartphone. HRV means were stratified by alcohol and IPV status at the prior report. Higher levels of HRV/Respiratory Sinus Arrhythmia represent better autonomic balance and physiological reactivity and low levels would represent more maladaptive physiological reactivity and autonomic imbalance.
Time Frame: From enrollment through end of evaluation period; 28 days.
Population: Analysis completed on N=83 participants who had at least one valid Heart Rate Variability measurement. N=9 participant were not included in the sample. N=2 lost to follow up. N=2 withdrew from the study. N=2 withdrawn by principal investigator. N=3 heart rate variability was not collected. The means below represent instances where reports were generated in each condition (e.g. HRV diary report when responder indicated no alcohol and no IPV)
Measure: Mean (Standard Deviation); unit: Milliseconds
Groups:
- Full Sample: Participants were N=46 couples with current alcohol use disorder and recent physical intimate partner violence (IPV). All participants completed 28 days of ecological momentary assessment (EMA; 4 times daily plus optional event-driven reports) of alcohol use, couple conflict including IPV, and affect via smartphone.
Arm/Group | Full Sample
Number analyzed (Participants) | 83
Milliseconds
  HRV/RSA Reports of No Alcohol and No Intimate Partner Violence (of 83 participants analyzed). | 58.60 (21.27)
  HRV/RSA Reports of No Alcohol and Yes Intimate Partner Violence (of 83 participants analyzed). | 62.28 (22.79)
  HRV/RSA Reports of Yes Alcohol and No Intimate Partner Violence (of 83 participants analyzed). | 59.32 (20.35)
  HRV/RSA Reports of Yes Alcohol and Yes Intimate Partner Violence (of 83 participants analyzed). | 60.15 (17.13)

2. Primary Outcome: Usability of Heart Rate Variability-Biofeedback Intervention
Description: Usability is assessed by the score on the self-report Post-Study System Usability Questionnaire (PSSUQ), ranging from 18-126. A low score indicates high usability of the Heart Rate Variability-Biofeedback (HRV-B) intervention, and a high score indicates low usability of the HRV-B intervention. Participants explore the device/app for 28 days and add the biofeedback technique for the final 7 days. They are asked to complete the PSSUQ during their exit interview.
Time Frame: During the exit interview, following 28 days of ecological momentary assessment (EMA).
Population: Participants analyzed include all participants who completed the Post-Study System Usability Questionnaire.
  Although N=86 participants completed the PSSUQ, one person responded with 'N/A' to all of the questions, thus creating an invalid response. Data was analyzed on N=85 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Total Sample: Participants were N=46 couples with current alcohol use disorder and recent physical intimate partner violence (IPV). All participants completed 28 days of ecological momentary assessment (EMA; 4 times daily plus optional event-driven reports) of alcohol use, couple conflict including IPV, and affect via smartphone.
Arm/Group | Total Sample
Number analyzed (Participants) | 85
score on a scale | 51.6 (23.7)

3. Primary Outcome: Feasibility of Heart Rate Variability-Biofeedback Intervention
Description: Feasibility is assessed by the rates of Heart Rate Variability-Biofeedback (HRV-B) task completion over the final 7 days. Higher rates of completion would indicate high feasibility of the Heart Rate Variability-Biofeedback (HRV-B) intervention, and low rates of completion would indicate low feasibility of the HRV-B intervention.
Time Frame: From days 21-28 during the Heart Rate Variability-Biofeedback (HRV-B) intervention; 7 days.
Population: Analysis completed on all 92 participants with Heart Rate Variability-Biofeedback data.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Sample
Number analyzed (Participants) | 92
Participants
  Completed intervention at least once | 78
  Completed intervention for at least 7 days | 21
  Completed 10 minutes of intervention for 7 days | 0

4. Primary Outcome: Acceptability of Heart Rate Variability-Biofeedback Intervention
Description: Acceptability is assessed by the score on the self-report measure Client Satisfaction Questionnaire (CSQ). Scores range from 8-32. A high score indicates high acceptability of the Heart Rate Variability-Biofeedback (HRV-B) intervention, and a low score indicates low acceptability of the HRV-B intervention. Participants explore the device/app for 28 days and add the biofeedback technique for the final 7 days. They are asked to complete the CSQ during their exit interview.
Time Frame: During the exit interview, following 28 days of ecological momentary assessment (EMA).
Population: Analysis completed on 86 participants with valid self report and Heart Rate Variability-Biofeedback data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total Sample
Number analyzed (Participants) | 86
score on a scale | 24.6 (5.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the course of the study (from baseline through the 28 day assessment period and the exit interview).
Groups:
- Total Sample: Participants were N=46 couples with current AUD and recent physical IPV. All participants completed 28 days of ecological momentary assessment (EMA; 4 times daily plus optional event-driven reports) of alcohol use, couple conflict including IPV, and affect via smartphone.
Arm/Group | Total Sample
All-Cause Mortality (participants affected / at risk) | 0/92
Serious Adverse Events (participants affected / at risk) | 0/92
Other Adverse Events (participants affected / at risk) | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT05374798/Prot_SAP_001.pdf
  • Informed Consent Form (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT05374798/ICF_000.pdf